CLINICAL TRIAL: NCT03133832
Title: Efficacy of Chinese-made Versus WHO-PQ Praziquantel for Treatment of Schistosoma Haematobium in Zanzibar: a Randomized Controlled Trial
Brief Title: The Chinese-made Praziquantel for Treatment of Schistosoma Haematobium
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Institute of Parasitic Diseases (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, YANG KUN, Deputy director, Jiangsu Institute of Parasitic Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIPD2017001
Record Dates: First submitted 2017-04-19; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Schistosomiasis Haematobia
Keywords: Schistosomiasis haematobium; Praziquantel; A randomized controlled trial
MeSH Terms: conditions — Schistosomiasis haematobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The cure rate between the two treatment (Experimental): Compare the cure rate between the Chinese-made praziquantel and companion tablet at one dose of 40 mg/kg
  Interventions: Drug: Companion Tablet
- The amount of eggs produced (Experimental): Compare the amount of eggs produced between the Chinese-made praziquantel and companion tablet at one dose of 40 mg/kg
  Interventions: Drug: Companion Tablet
- The economic benefit (Experimental): Compare the economic benefit between the Chinese-made praziquantel and companion tablet at one dose of 40 mg/kg
  Interventions: Drug: Companion Tablet

INTERVENTIONS:
Drug: Companion Tablet — Chinese-made drug for schistosomiasis treatment
  Other Names: Chinese-made praziquantel

SUMMARY:
Schistosomiasis remains an important parasitic disease in the tropics, special in Africa including Zanzibar. The WHO-recommended strategy to eliminate schistosomiasis involves large-scale treatment of affected populations through periodic, targeted treatment of school-children with praziquantel. Donated praziquantel is the key to achieving elimination. The increase in the number of treatments is attributable to many factors, including improved availability of donated praziquantel, essentially from Merck; new countries starting to implement large-scale schistosomiasis control programmes; geographical scale-up of treatment within countries; and improved reporting to WHO. The global target set by WHO in the Roadmap on neglected tropical diseases is to attain at least 75% coverage of preventive chemotherapy in pre-school and school-age children by 2020. Experience from China demonstrates that preventive chemotherapy (that is, large scale treatment without individual diagnosis) with high coverage can significantly impact indices of infection and reduce transmission. The praziquantel made in China has been used from 1990s, and have effectively activity against S. haematobium, special the good economic benefits.

The project will propose to conduct an open-label, randomized trial to evaluate the comparative efficacy of Chinese-made Praziquantel versus WHO Praziquantel in the treatment of 200 people infected with S. haematobium in Pemba island Zanzibar. To do this the investigators will screen about 4000 people by examination of urine for schistosome eggs. Eligible participants will be randomized to receive a single dose of Chinese-made and WHO Praziquantel. Four weeks after treatment, the participants will be assessed for cure and egg reduction. The study may provide an alternative drug treatment for S. haematobium.

DETAILED DESCRIPTION:
Participants There about 4000 peoples (aged 7-60 years) were enrolled from three Shehias in Pemba island Zanzibar. Urine will be collected and tested on April 2017. Eligible people will be enrolled based on the criteria of inclusion and exclusion. A series of meetings will be held at Shehias and schools to explain the objectives, procedures, and potential risks of the study.

Randomization Participants were randomly assigned (1:1) to receive Chinese-made versus WHO-PQ praziquantel. The randomization sequence was computer generated by the study sponsor. The staff of NTD office will give the assigned study drug after confirming the treatment allocation from the randomisation sequence. The NTD staff and and study participants will be unmasked to treatment assignment, but the laboratory technicians will be masked to treatment assignment throughout the study.

Procedures Firstly, every participant provided a fresh urine sample, which was used to detect the presence of S. haematobium. The NTD staff will do a physical examination, and checked the eligibility of every participant.

Participants whose urines tested positive for S. haematobium eggs and who met all eligibility criteria were invited to participate in the study.

Chines-made and WHO-PQ praziquantel will be give the participants one dose of 40 mg/kg per day. All study drugs were given orally, and the NTD staff will also record the exact time of drug ingestion.

Participants will be observed for 2 h after taking the drug to ensure retention and check for any immediate adverse events. If vomiting occurred within 2 h of drug ingestion, a second full dose was given.

After one month after enrolment, the follow-up visit will be provided, and urine will be collected and tested for S. haematobium eggs. As a quality control measure for inter-observer variability, a third technician reread a random selection of 10% of slides.

An adverse event is defined as a sign, symptom, intercurrent illness, or abnormal laboratory finding that just occurred during follow-up.

At the end of the study, all participants who have still excreting S. haematobium eggs (ie, not cured) will be treated with praziquantel again.

Statistical analysis There serial report forms will be used to data collection from participants, and Epi Info will be used to data enter.

The cure rate, the mean egg count and economic benefits will be analysed between the different group.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 7 and 60 years old
* Study participants appear healthy at enrollment
* Suffering from S. haematobium infection, excreting eggs in urine
* Residing in Pemba island, Zanzibar
* Able to receive oral treatment
* Assent to participate in study

Exclusion Criteria:

* Pregnant or lactating at the time of the study
* Presence of severe illness or malnutrition
* Hypersensitivity to PZQ.

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-07-10 (Estimated)

PRIMARY OUTCOMES:
The cure rate of the two treatment | After one month
  Collect urines from all participants for the group of Chinese-made and WHO-PQ praziquantel, test in the laboratory, calculate the proportion of patients cured, namely, the the cure rate. And then compare the cure rate between Chinese-made and WHO-PQ praziquantel.

SECONDARY OUTCOMES:
The egg reduction of the two treatment | After one month
  Collect urines from all participants for the group of Chinese-made and WHO-PQ praziquantel, test in the laboratory, get the account of eggs of each particpant, calculate the proportion of excreting S. haematobium eggs, and the egg reduction rate. And then compare the gg reduction rate between Chinese-made and WHO-PQ praziquantel.

OTHER OUTCOMES:
The economic benefit of the two treatment | After one and half month
  Collect questionnaires from all participants for the group of Chinese-made and WHO-PQ praziquantel, including the side effects, the cost of tables and deliver etc. And then compare the economic benefit between Chinese-made and WHO-PQ praziquantel.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Yang, PHD, Principal Investigator — Jiangsu Institute of Parasitic Diseases
Locations (1):
- NTD office, Pemba,Ministry of Health, Zanzibar, Pemba, Zanzibar, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang XY, He J, Juma S, Kabole F, Guo JG, Dai JR, Li W, Yang K. Efficacy of China-made praziquantel for treatment of Schistosomiasis haematobium in Africa: A randomized controlled trial. PLoS Negl Trop Dis. 2019 Apr 10;13(4):e0007238. doi: 10.1371/journal.pntd.0007238. eCollection 2019 Apr. PMID 30969960